CLINICAL TRIAL: NCT03694145
Title: Predicting Diabetic Retinopathy From Risk Factor Data and Digital Retinal Images
Status: Active, not recruiting | Type: Observational
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Library of Medicine (NLM) (NIH); Los Angeles County Department of Public Health (Other Government); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 1218589-3; R01LM012309 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients w. risk of retinopathy: The 300-500 patients to be enrolled for the study are diabetic patients normally seen by the Los Angeles County Department of Health Services (LACDHS) Teleretinal Diabetic Retinopathy Screening Program and Reading Center. In addition to receiving their recommended LACDHS annual teleretinal screening, for the study, participants will receive an additional in-person eye examination.
  Interventions: Other: In-Person Eye Examination

INTERVENTIONS:
Other: In-Person Eye Examination — Dilated in-person eye examination by a board-certified ophthalmologist or retinal fellow.

SUMMARY:
The objective of this study is to compare the results of a deep learning approach to diabetic retinopathy assessment with results from (1) an in-person examination with an ophthalmologist, and (2) the assessments of optometrists involved in a teleretinal screening program.

DETAILED DESCRIPTION:
This study represents the third aim of a grant with five aims. The study will compare and evaluate the predictive accuracy of: (a) machine learning models developed to grade diabetic retinopathy and assess the presence or absence of diabetic macular edema and (b) the assessments of optometrist readers, both from digital retinal images, against standard of care dilated retinal examinations by board-certified ophthalmologists and/or retinal-specialty fellows for 300 diabetic patients utilizing a Los Angeles County reading center.

For the study, the investigators will recruit 300-500 eligible diabetic patients for in-person eye examinations performed by board certified ophthalmologists and/or retinal-specialty fellows at Los Angeles County reading centers. The study will take place over the course of two visits: a teleretinal screening and an in-person eye examination.

The in-person dilated eye examinations that the study participants will participate in and be compensated for follow the usual standard of care that patients receive in a setting that does not utilize teleretinal screening. Yearly dilated eye examinations are standard of care for all persons with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Type I or Type II Diabetes
* Patients who are over the age of 18 years
* Patients who have not previously been seen in the current year by the LACDHS Teleretinal Diabetic Retinopathy Screening Program and Reading Center
* Patients whose teleretinal screening exam images yield readable results

Exclusion Criteria:

* Patients under the age of 18 years
* Patients with gestational diabetes
* Patients who have previously been seen in the current year by LACDHS's Teleretinal Diabetic Retinopathy Screening Program and Reading Center
* Patients whose teleretinal screening exam images do not yield readable results, as gradable images are needed for later comparison against ophthalmologist reads.
* Previously eligible patients who do not return for an in-person eye exam within 3 months of receiving a teleretinal screening (In order for the results of the teleretinal screening and in-person eye examinations to yield similar information, patients who do not return for their in-person eye exam within 3 months of their teleretinal screening will not be able to remain in the study. This is because significant eye changes not documented by the teleretinal screening may occur after a 3-month period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients with Type I or Type II diabetes who are normally seen at LACDHS clinics and usually screened for diabetic retinopathy via teleretinal screening.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients accurately diagnosed with retinopathy | 11/2022
  Proportion of patients accurately diagnosed with retinopathy using machine learning versus proportion accurately diagnosed by teleretinal screening optometrists with in-person eye examinations by ophthalmologists used as a gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Omolola Ogunyemi, PhD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (3):
- United States (3):
  - Los Angeles Department of Public Health, Los Angeles, California
  - University of California - Los Angeles, Los Angeles, California
  - Charles R. Drew University of Medicine and Science, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No